CLINICAL TRIAL: NCT02279368
Title: Nursing Led Interdisciplinary Intervention in Prevention of Girl Child Mortality and Maltreatment: Randomized Controlled Trial
Brief Title: Nursing Led Interdisciplinary Intervention in Prevention of Girl Child Mortality and Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adwin Life Care (Industry)
Collaborators: Sonal Foundation, India (Other); Gyaansanjeevani, Jhunjhunu, Rajasthan, India (Unknown); Khatri education trust, Satnaali, Hariyana, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Adwin006
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Abuse Neglect Social; Deprivation, Maltreatment Syndrome (Infant or Child)
MeSH Terms: interventions — Family Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Nurses delivered the supportive intervention along with family counselling from last term of pregnancy through three months and then were followed till the first birthday of the child.
  Interventions: Behavioral: Family Counselling and safeguarding
- Control Group (No Intervention): Control group families were followed in usual care.

INTERVENTIONS:
Behavioral: Family Counselling and safeguarding
  Arms: Intervention Group

SUMMARY:
In Northern India, skewed sex ratios, female feticide and higher child mortality rates for girls have become serious concern. The female child mortality as a result of son preference have increased during the last several decades. Since families cannot know the sex of the fetus due to Indian government policies, they now 'neglect' girl child to ensure there are few survivors. Survival chances of second and third daughters are plunging neglecting healthcare and nutrition has become tool for death as 'good riddance'.

ELIGIBILITY:
Inclusion Criteria:

* Families having girl child before
* High risk families with high expectation of having son

Exclusion Criteria:

* Families having son before
* Relocation and moving out of town during study period
* Not ready to consent for intervention

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mother-infant interaction (Parent/Caregiver Involvement Scale) | Change from Baseline in Parent/Caregiver Involvement Scale at 6 weeks

SECONDARY OUTCOMES:
Abuse and neglect outcomes (reported incidences of abuse and maltreatment) | Upto six weeks reported incidences of abuse and maltreatment

OTHER OUTCOMES:
Child survival rate (reported incidences of injuries and emergencies) | Upto six weeks reported incidences of injuries and emergencies

CONTACTS AND LOCATIONS:
Overall Officials: Alpesh Barot, MA, Principal Investigator — Sonal Foundation, India; Valerie Murray, MA, Study Director — Macmillan Research Group
Locations (3):
- India (3):
  - Sonal Foundation, Mahesāna, Gujarat
  - Khatri educational trust, Satnāli, Haryana
  - GyanSanjeevani, Jhunjhunūn, Rajasthan